CLINICAL TRIAL: NCT03966027
Title: Immediate Vs. Delayed Weight Bearing Postoperative Protocol in Diabetic Ankle Fractures
Acronym: Diabetic Ankle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Schweser MD (Other)
Responsible Party: Sponsor-Investigator, Kyle Schweser MD, Assistant Professor Orthopaedic Trauma/Foot and Ankle, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014997
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ankle Fractures
Keywords: Diabetic Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: Diabetic patients with ankle fractures will be manage operatively and then randomized to be prescribed a hindfoot offloading brace 2 weeks after surgery or be randomized to follow a non-immediate weight bearing rehabilitation protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hindfoot Offloading Braces / Immediate Weight-bearing (Experimental): Diabetic patients over 18 years of age who sustained an isolated (non-pilon) ankle fracture will undergo ORIF of the ankle fracture within 3 weeks of the event
  Interventions: Other: Postoperative protocol (Immediate weight bearing)
- No Hindfoot Offloading Braces / Delayed Weight-Bearing (Placebo Comparator): Diabetic patients over 18 years of age who sustained an isolated (non-pilon) ankle fracture will undergo ORIF of the ankle fracture within 3 weeks of the event
  Interventions: Other: Postoperative Protocol (Delayed Weight Bearing)

INTERVENTIONS:
Other: Postoperative protocol (Immediate weight bearing) — After ORIF of the ankle fracture, the patient will be randomized to follow an immediate weight bearing rehabilitation protocol using an offloading hindfoot brace
  Arms: Hindfoot Offloading Braces / Immediate Weight-bearing
Other: Postoperative Protocol (Delayed Weight Bearing) — After ORIF of the ankle fracture, the patient will be randomized to follow a standard delayed weight-bearing rehabilitation protocol
  Arms: No Hindfoot Offloading Braces / Delayed Weight-Bearing

SUMMARY:
Operatively managed diabetic ankle fractures have significant risk for complications. The cause for failure is likely multifactorial, however, a component of failure has to do with an inability to process pain and pressure normally. This loss of protective sensation allows for an increase in abnormal stresses placed on the recently repaired fractures. Historically, diabetics have been kept non weight bearing for extended periods of time, which has its own functional and cardiovascular issues. The purpose of the study is to determine if a protocol of immediate weight bearing with a hindfoot offloading brace after surgically corrected ankle fracture in a diabetic patient will maintain adequate motion, have no difference in complications when compared to regular non-immediate weight bearing protocols, and lead to good outcome scores and patient satisfaction scores

DETAILED DESCRIPTION:
Operatively managed diabetic ankle fractures have significant risk for complications. The cause for failure is likely multifactorial, however, a component of failure has to do with an inability to process pain and pressure normally. This loss of protective sensation allows for an increase in abnormal stresses placed on the recently repaired fractures. Historically, diabetics have been kept non weight bearing for extended periods of time, which has its own functional and cardiovascular issues. The purpose of the study is to determine if a protocol of immediate weight bearing with a hindfoot offloading brace after surgically corrected ankle fracture in a diabetic patient will maintain adequate motion, have no difference in complications when compared to regular non-immediate weight bearing protocols, and lead to good outcome scores and patient satisfaction scores

Patients will be recruited from the trauma and foot & ankle service lines. Patients who have experienced an isolated ankle fracture (excluding pilon fracture) and will undergo operative fixation within 3 weeks of injury will be approached for consent. Patients will then be screened based on the inclusion and exclusion criteria. Up to 25 patients will be enrolled

The following protocol will be applied after enrollment

1. Pre-operatively

   a. Hemoglobin A1c will also be collected from each patient if it has not been performed within the last 30 days.
2. Post-operatively a. Post-surgery i. Standard of Care:

1. Placement into short leg, non-weight bearing splint to allow for wound healing and brace fabrication ii. Research Specific:

1. Fitted for brace (will be custom made and take approximately 1-2 weeks) b. 2 week visit (standard of care timepoint) i. Standard of Care:

1. Placed into compression stockings
2. Counseling regarding skin checks and diabetic skin care
3. Physical therapy prescription given ii. Research Specific

1. Placement into brace so it offloads the hindfoot to 15 pounds of pressure or less 2. Education by prosthetist, physiatrist, and/or attending physician about proper brace wear and maintenance, and the importance of weight bearing only in brace.

c. 3 Week visit (not standard of care timepoint) i. Research Specific

1. Ankle radiographs d. 4 weeks, 6 weeks, 12 Weeks, 26 weeks, and 1 year visits (standard of care time points) i. Standard of Care

1. Surveys (PROMIS, AAOS Foot and Ankle)
2. Ankle Radiographs ii. Research Specific

1. Counseling regarding brace wear 2. Brace adjustments as needed e. 8 week, 10 week, 14 week, 16 week, (non-standard of care biweekly visits until healing occurs) i. Research Specific

1. Ankle Radiographs (if early failure is suspected)
2. Skin Check

Upon study completion, patients will continue with post-operative rehab following the surgeon's standard of care. If a patients is removed prematurely or if the study ends prematurely, they will receive standard of care procedures going forward

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 and ove
2. Positive for diabetes
3. Positive monofilament test
4. Isolated ankle fracture (non-pilon) and undergoing operative intervention within 3 weeks of fracture
5. Weight less than 275 (124kg)
6. Can tolerate and comply with brace
7. No signs of pre-existing charcot arthroplasty or ankle deformity

Exclusion Criteria:

1. Children
2. Pregnant patients
3. No signs of diabetes complicated by neuropathy
4. Non-operative ankle fractures
5. Multiple extremity injury
6. Cannot follow post-operative protocol
7. Chronic ankle fractures receiving surgery beyond 3 weeks of injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Adverse Events by type over time, severity, seriousness, and relatedness. AEs will be tabulated and summarized as counts and percentages. AEs will also be cross-tabulated according to:
  1. Severity;
  2. Unanticipated Adverse Device Effect (UADE)
  3. Seriousness (Serious Adverse Event (SAE), Non-serious AE);
  4. Device-Relatedness (Unrelated, Possibly Related, Probably Related, Definitely Related);
  5. Procedure-Relatedness (Unrelated, Possibly Related, Probably Related, Definitely Related).

SECONDARY OUTCOMES:
AAOS Foot and Ankle Score | 12 Months
  The AAOS foot and ankle questionnaire is a patient-administrated 25-item survey specifically developed for foot and ankle-related disability. The questionnaire is divided into two scales, the Foot and Ankle Core scale, comprised of 20 questions and the Shoe Comfort Scale with five questions. The questions themselves are distributed among five different categories: Pain (9 items), function (6 items), stiffness and swelling (2 items), giving way (3 items) and shoe comfort (5 items). Answers are then measured on a scale of 1 to 5 or 6, with 1 being the best outcome score.
PROMIS Score | 12 Months
  The Patient-Reported Outcomes Measurement Information System® (PROMIS) is a flexible set of tools designed to measure self-reported physical, mental and social health and wellbeing. PROMIS instruments contain a fixed number of items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The questionarie assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. Norm-based scores are calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population (standard deviation = 10).

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Schweser, MD, Principal Investigator — Assistant Professor Orthopaedic Trauma/Foot and Ankle
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The Investigator will maintain all study records according to applicable University regulatory requirement(s). Hard copy records will be retained for at least 7 years after the last clinic follow-up visit at the Missouri Orthopaedic Institute in a locked filing cabinet. Electronic records will be retained for the same amount of time but on secured computers and servers. If the Investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility.

REFERENCES:
- [Background] Raghav A, Khan ZA, Labala RK, Ahmad J, Noor S, Mishra BK. Financial burden of diabetic foot ulcers to world: a progressive topic to discuss always. Ther Adv Endocrinol Metab. 2018 Jan;9(1):29-31. doi: 10.1177/2042018817744513. Epub 2017 Dec 12. PMID 29344337
- [Background] Jani MM, Ricci WM, Borrelli J Jr, Barrett SE, Johnson JE. A protocol for treatment of unstable ankle fractures using transarticular fixation in patients with diabetes mellitus and loss of protective sensibility. Foot Ankle Int. 2003 Nov;24(11):838-44. doi: 10.1177/107110070302401106. PMID 14655888
- [Background] Shehab DK, Al-Jarallah KF, Abraham M, Mojiminiyi OA, Al-Mohamedy H, Abdella NA. Back to basics: ankle reflex in the evaluation of peripheral neuropathy in type 2 diabetes mellitus. QJM. 2012 Apr;105(4):315-20. doi: 10.1093/qjmed/hcr212. Epub 2011 Nov 8. PMID 22071964
- [Result] Wukich DK, Kline AJ. The management of ankle fractures in patients with diabetes. J Bone Joint Surg Am. 2008 Jul;90(7):1570-8. doi: 10.2106/JBJS.G.01673. PMID 18594108
- [Result] Holder CG, Haskvitz EM, Weltman A. The effects of assistive devices on the oxygen cost, cardiovascular stress, and perception of nonweight-bearing ambulation. J Orthop Sports Phys Ther. 1993 Oct;18(4):537-42. doi: 10.2519/jospt.1993.18.4.537. PMID 8220412